CLINICAL TRIAL: NCT03811353
Title: Reliability and Validity of the Turkish Mastication Observation and Evaluation (T-MOE) Instrument
Brief Title: The Turkish Mastication Observation and Evaluation (T-MOE) Instrument
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: ArslanSerel2019
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Chewing Problem; Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with cerebral palsy: Chewing performance will be evaluated with T-MOE and the Karaduman Chewing Performance Scale. Tongue control will also be evaluated by Tongue Thrust Rating Scale.
  Interventions: Diagnostic Test: T-MOE
- Healthy children: Chewing performance will be evaluated with T-MOE and the Karaduman Chewing Performance Scale. Tongue control will also be evaluated by Tongue Thrust Rating Scale.
  Interventions: Diagnostic Test: T-MOE

INTERVENTIONS:
Diagnostic Test: T-MOE — Chewing performance will be evaluated with T-MOE and the Karaduman Chewing Performance Scale.

SUMMARY:
The purpose of this study is to test the reliability and validity of the T-MOE among pediatric patients with chewing disorders.

DETAILED DESCRIPTION:
The purpose of this study is to test the reliability and validity of the T-MOE among pediatric patients with chewing disorders.The internal consistency, test-retest reliability, and criterion validity of T-MOE will be investigated. The internal consistency will be assessed using Cronbach's alpha. Intraclass correlation coefficient (ICC) value with 95 % confidence intervals will be calculated for test-retest reliability. The criterion validity of the scale will be determined by assessing the correlation between the T-MOE and Karaduman Chewing Performance Scale and Tongue Thrust Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Having chewing disorders aged between 18 months-12 years
* Being serebral palsy
* Being healthy children

Exclusion Criteria:

* No chewing disorders
* A child aged below 6 months

Ages: 18 Months to 12 Years | Sex: All
Age Groups: Child
Study Population: Children with serebral palsy and healthy children
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
The Turkish Mastication Observation and Evaluation (T-MOE) Instrument | 3 months
  This instrument is used to evaluate chewing function in children. The T-MOE includes 8 items, and could be scored between 1 to 4. Higher scores indicate better chewing function, lower scores indicate worse chewing function.

SECONDARY OUTCOMES:
The Karaduman Chewing Performance Scale (KCPS) | 3 months
  This scale is used to determine chewing performance level of children. The KCPS has 5 steps including 0 to 4. 0 means 'Normal chewing function' and 4 means 'No biting and chewing'.
Tongue Thrust Rating Scale (TTRS) | 3 months
  This scale is used to determine tongue thrust severity of children. The TTRS has 4 steps between 0 to 3. Step 0 means 'No tongue thrust.' and step 3 means 'Severe tongue thrust. The tongue is positioned out of the mouth.'

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serel Arslan S, Demir N, Karaduman AA. Turkish Version of the Mastication Observation and Evaluation (MOE) Instrument: A Reliability and Validity Study in Children. Dysphagia. 2020 Apr;35(2):328-333. doi: 10.1007/s00455-019-10035-8. Epub 2019 Jul 10. PMID 31292728